CLINICAL TRIAL: NCT00765648
Title: A Phase IV, Randomized Trial to Determine the Efficacy and Safety of Cardene Intravenous (I.V.) Versus Labetalol for Management of Hypertensive Emergencies in the Emergency Department Setting
Brief Title: Evaluation of Intravenous Cardene(Nicardipine)and Labetalol Use in the Emergency Department
Acronym: CLUE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: EKR Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-001
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2011-07

CONDITIONS: Hypertensive Urgency
Keywords: hypertension; emergency department; Nicardipine; Labetalol; hypertensive emergency; hypertensive urgency
MeSH Terms: conditions — Hypertensive Crisis; Hypertension; Emergencies | interventions — Nicardipine; Labetalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): nicardipine intravenous
  Interventions: Drug: nicardipine intravenous
- 2 (Active Comparator): Labetalol
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: nicardipine intravenous — nicardipine intravenous 5 mg/hour titrated every 5 minutes by 2.5 mg/hour until target systolic blood pressure range (TSBPR) is reached or maximum dose of 15 mg/hour is achieved.Following achievement of target systolic blood pressure range the infusion rate should be decreased to 3 mg/hour
  Other Names: Nicardipine hydrochloride
  Arms: 1
Drug: Labetalol — Labetalol: bolus therapy to start at 20 mg intravenous injection over 2 minutes, may repeat 20mg, 40mg or 80mg injections every 10 minutes until target systolic blood pressure range(TSBPR)is reached or a maximum of 300 mg is injected.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Cardene I.V. to labetalol administered intravenously for the management of hypertension in the emergency department setting.

DETAILED DESCRIPTION:
More than 3 million patients yearly receive an intravenous antihypertensive agent in the US. Despite this large number of critically ill patients treated annually, little research exists in the area of acute severe hypertension, specifically hypertensive emergency, a serious condition that contributes to morbidity and mortality.

Two agents that are commonly used to treat acute hypertensive crisis include labetalol and nicardipine. Cardene may provide benefits in titration and has shown to have lower dosage adjustments compared to labetalol. Nicardipine has also shown a decreased need for additional antihypertensives when compared to labetalol in patients with stroke in a neurological ICU.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Systolic blood pressure ≥180 mm Hg on 2 consecutive readings(10 minutes apart)presenting in the emergency department (ED)

Exclusion Criteria:

* Use of any investigational drug within 1 month prior to emergency department (ED)
* Pregnant or breast-feeding females
* Contraindications or allergy to beta-blockers and calcium channel blockers (see FDA approved labeling for nicardipine intravenous and labetalol)
* Subjects with decompensated congestive heart failure (CHF) or with a known left ventricular ejection fraction (LVEF) <35%
* History of stroke within 30 days
* Known liver failure
* Suspected myocardial infarction
* Suspected aortic dissection
* Suspected cocaine overdose
* Concurrently receiving other intravenous (I.V.) hypertensive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Frank Peacock, MD, Principal Investigator — The Cleveland Clinic; Joseph Varon, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Health Science Center, Houston, Texas

REFERENCES:
- [Derived] Varon J, Soto-Ruiz KM, Baumann BM, Borczuk P, Cannon CM, Chandra A, Cline DM, Diercks DB, Hiestand B, Hsu A, Jois-Bilowich P, Kaminski B, Levy P, Nowak RM, Schrock JW, Peacock WF. The management of acute hypertension in patients with renal dysfunction: labetalol or nicardipine? Postgrad Med. 2014 Jul;126(4):124-30. doi: 10.3810/pgm.2014.07.2790. PMID 25141250
- [Derived] Cannon CM, Levy P, Baumann BM, Borczuk P, Chandra A, Cline DM, Diercks DB, Hiestand B, Hsu A, Jois P, Kaminski B, Nowak RM, Schrock JW, Varon J, Peacock WF. Intravenous nicardipine and labetalol use in hypertensive patients with signs or symptoms suggestive of end-organ damage in the emergency department: a subgroup analysis of the CLUE trial. BMJ Open. 2013 Mar 26;3(3):e002338. doi: 10.1136/bmjopen-2012-002338. PMID 23535700
- [Derived] Peacock WF, Varon J, Baumann BM, Borczuk P, Cannon CM, Chandra A, Cline DM, Diercks D, Hiestand B, Hsu A, Jois-Bilowich P, Kaminski B, Levy P, Nowak RM, Schrock JW. CLUE: a randomized comparative effectiveness trial of IV nicardipine versus labetalol use in the emergency department. Crit Care. 2011;15(3):R157. doi: 10.1186/cc10289. Epub 2011 Jun 27. PMID 21707983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients had 2 systolic blood pressures(BP) measures > 180 mmHg at least 10 minutes apart, and no contraindications.Emergency room setting.
Groups:
- Nicardipine Dosing Was 5 mg/Hour: nicardipine intravenous
- Bolus Labetalol Began at 20 mg Over 2 Minutes: Labetalol
Period: Overall Study
Arm/Group | Nicardipine Dosing Was 5 mg/Hour | Bolus Labetalol Began at 20 mg Over 2 Minutes
Started | 110 | 116
Completed | 109 | 114
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicardipine Dosing Was 5 mg/Hour | Bolus Labetalol Began at 20 mg Over 2 Minutes | Total
Number analyzed (Participants) | 110 | 116 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 98 | 179
  >=65 years | 29 | 18 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 59 | 119
  Male | 50 | 57 | 107
Region of Enrollment [Number; unit: participants]
  United States | 110 | 116 | 226

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving a Pre-defined Target Systolic Blood Pressure (BP) Within 30 Minutes.
Description: Percentage of subjects achieving a pre-defined target systolic blood pressure (BP) range defined as a systolic blood pressure that is within +/- 20 mmHg of the target as established by the investigator.
Time Frame: 30 minutes after initiation of therapy
Population: Intent to treat cohort.
Measure: Number; unit: percentage of participants
Groups:
- Nicardipine: Nicardipine was administered at 5mg/hour and increased every 5 minutes by 2.5 mg/hour until the target systolic blood pressure (SBP) range is reached or maximum of 15mg/hour is achieved.
- Labetalol: Labetalol is given intravenous bolus starting with 20mg over 2 minutes, which is repeated at 20, 40, or 80mg injections every 10 minutes until the target systolic blood pressure (SBP) range is reached or a maximum of 300mg is administered.
Arm/Group | Nicardipine | Labetalol
Number analyzed (Participants) | 109 | 114
percentage of participants | 91.7 | 82.5
Statistical Analysis 1: Comparison: Nicardipine vs Labetalol; Test type: Superiority or Other; p = 0.04, Chi-squared; Risk Difference (RD) = -9.3, 95% CI 2-sided [-18.0 to -0.6]

2. Secondary Outcome: Average Number of Dose Titrations Within 30 Minutes
Description: Calculated as the mean (± standard deviation) number of titrations over 30 minutes for each treatment group
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: number of titrations
Arm/Group | Nicardipine | Labetalol
Number analyzed (Participants) | 109 | 114
number of titrations | 2.2 (1) | 1.3 (0.97)
Statistical Analysis 1: Comparison: Nicardipine vs Labetalol; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Emergency Department(ED)Time to Disposition Decision
Description: Median number of hours from hospital admission until Emergency Department(ED)disposition
Time Frame: 6 hours
Population: these are the correct participant numbers for this secondary analysis
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nicardipine | Labetalol
Number analyzed (Participants) | 109 | 115
hours | 4.6 [3.5 to 6.6] | 4.6 [3.1 to 7.6]
Statistical Analysis 1: Comparison: Nicardipine vs Labetalol; Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Treatment Failure
Description: Treatment failure is defined as admission to the hospital or observation unit for BP management
Time Frame: 6 hours
Population: these are the correct participant numbers for this secondary analysis
Measure: Number; unit: percentage of participants
Arm/Group | Nicardipine | Labetalol
Number analyzed (Participants) | 109 | 115
percentage of participants | 43.1 | 37.4
Statistical Analysis 1: Comparison: Nicardipine vs Labetalol; Test type: Superiority or Other; p = 0.38, Chi-squared

5. Secondary Outcome: Subjects Requiring the Use of Intravenous Rescue Medications
Description: The percent of subjects requiring the use of intravenous rescue medications
Time Frame: 6 hours
Measure: Number; unit: percentage of participants
Arm/Group | Nicardipine | Labetalol
Number analyzed (Participants) | 110 | 116
percentage of participants | 15.5 | 22.4
Statistical Analysis 1: Comparison: Nicardipine vs Labetalol; Test type: Superiority or Other; p = 0.18, Chi-squared

6. Secondary Outcome: Transition Time to Oral Medication
Description: The median transition time (in hours) to oral medication
Time Frame: 6 hours
Population: these are the correct participant numbers for this secondary analysis
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nicardipine | Labetalol
Number analyzed (Participants) | 96 | 85
hours | 4.9 [1.4 to 10.9] | 6.4 [2.2 to 16.5]
Statistical Analysis 1: Comparison: Nicardipine vs Labetalol; Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Emergency Room visit
Description: Elevated cardiac markers
Groups:
- Nicardipine: Nicardipine dosing was 5 mg/hour
- Labetalol: Bolus Labetalol began at 20 mg over 2 minutes
Arm/Group | Nicardipine | Labetalol
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/116
Other Adverse Events (participants affected / at risk) | 1/110 | 0/116
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicardipine (N=110) | Labetalol (N=116)
Elevated cardiac biomarkers (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less